CLINICAL TRIAL: NCT00004406
Title: Randomized Study of Human Parathyroid Hormone in Middle-Aged Men With Idiopathic Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13293; CPS-CU-FDR001024
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-01

CONDITIONS: Osteoporosis
Keywords: disease-related problem/condition; osteoporosis; rare disease
MeSH Terms: conditions — Osteoporosis; Rare Diseases | interventions — PTH protein, human

INTERVENTIONS:
Drug: human parathyroid hormone

SUMMARY:
OBJECTIVES:

I. Determine the effect of human parathyroid hormone (1-34) on bone mass in middle-aged men with idiopathic osteoporosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled study. All patients self-administer daily subcutaneous injections of human parathyroid hormone (1-34) or placebo for a period of 2.5 years.

Patients are followed regularly for unacceptable toxicities.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Osteoporosis as defined by: Bone mineral density at the lumbar spine or femoral neck that is 2.5 standard deviations below peak bone mass reference value (T score less than -2.5)

No family history of male osteoporosis

No other metabolic bone disease

--Prior/Concurrent Therapy--

Endocrine therapy:

* No concurrent glucocorticoid therapy
* No prior steroid use

Surgery: No prior gastrointestinal tract surgery

Other: No prior or concurrent anticonvulsant therapy

--Patient Characteristics--

Hematopoietic: Normal CBC

Hepatic: Normal liver function

Renal: Normal renal function

Other:

* Normal thyroid function
* Normal adrenal function
* Normal gonadal status
* No myeloma or other malignancy
* No alcoholism, hypercortisolism or diabetes mellitus
* No gastrointestinal tract disease or disorder associated with malabsorption

Ages: 29 Years to 67 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 1999-10; Study Completion 2004-07

CONTACTS AND LOCATIONS:
Overall Officials: John Paul Bilezikian, Study Chair — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States